CLINICAL TRIAL: NCT06369753
Title: Tratamiento de la distensión Abdominal Funcional
Brief Title: Visible Abdominal Distension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)459/2023B
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Irritable Bowel Syndrome; Dyspepsia; Functional Bloating
MeSH Terms: conditions — Irritable Bowel Syndrome; Dyspepsia | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Experimental)
  Interventions: Behavioral: Biofeedback
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Biofeedback — Three sessions of biofeedback intervention will be performed during the first 3 weeks of the intervention period. Patients will be taught to control abdominal and thoracic muscular activity by providing instructions using an original video support. Patients will be instructed to perform the same exercises before and after breakfast, lunch and dinner during the 4-week intervention period
  Arms: Biofeedback
Behavioral: Placebo — Three sessions of placebo intervention will be performed during the first 3 weeks of the intervention period. Sham measurements of abdominal and thoracic motion will be performed, and a pill of placebo containing 0.21 g glucose will be administered; patients will be instructed to take a pill of placebo before breakfast, lunch and dinner during the 4-week intervention period.
  Arms: Placebo

SUMMARY:
Background. Abdominal distention is produced by an abnormal somatic postural tone. The authors developed an original biofeedback technique. In a randomized, placebo-controlled trial the authors demonstrated the superiority of biofeedback over placebo for the treatment of abdominal distention. However, the technique is technically complex and unpractical.

Aim. To prove the efficacy of a noninstrumental biofeedback technique, transmitted by a standard training program, for the treatment of abdominal distension in different centers.

Selection criteria. Episodes of visible abdominal distension. Intervention. Patients will be randomized into biofeedback and placebo groups. Three sessions of either biofeedback or placebo intervention will be performed during the first 3 weeks of the intervention period.

Biofeedback: Patients will be taught to control abdominal and thoracic muscular activity by providing instructions using an original video support. In each center one operator will receive a standard training on how to deliver the noninstrumental biofeedback treatment. Patients will be instructed to perform the same exercises before and after breakfast, lunch and dinner during the 4-week intervention period.

Placebo: Sham measurements of abdominal and thoracic motion will be performed, and a pill of placebo containing 0.21 g glucose will be administered; patients will be instructed to take a pill of placebo before breakfast, lunch and dinner during the 4-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* episodes of visible abdominal distension triggered by meal ingestion

Exclusion Criteria:

* organic cause detected by clinical work-up
* constipation
* abdominal distension not confirmed by the 7-day clinical questionnaires in the pre- intervention evaluation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Visible abdominal distension | 4 weeks
  Distension score measured by scales graded from 0 (not at all) to 10 (very much) at the end of each day over a 7-day clinical evaluation period before and during the 4th week of the intervention.

SECONDARY OUTCOMES:
Sensation of abdominal pressure/fullness | 4 weeks
  Sensation score measured by scales graded from 0 (not at all) to 10 (very much) at the end of each day over a 7-day clinical evaluation period before and during the 4th week of the intervention.
Sensation of abdominal discomfort/pain | 4 weeks
  Sensation score measured by scales graded from 0 (not at all) to 10 (very much) at the end of each day over a 7-day clinical evaluation period before and during the 4th week of the intervention

OTHER OUTCOMES:
Follow-up after biofeedback | 6 months
  Sensation of abdominal distension measured by scales graded from 0 (not at all) to 10 (very much) at the end of each day over a 7-day clinical evaluation period at 1, 3 and 6 months after biofeedback treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Azpiroz, MD, Principal Investigator — University Hospital Vall d'Hebron
Locations (7):
- G. Oppenheimer Center for Neurobiology of Stress and Resilience, Los Angeles, California, United States
- McMaster University, Hamilton, Ontario, Canada
- Bordeaux University Hospital, Bordeaux, France
- Santa Orsola Hospital, Bologna, Italy
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- Sahlgrenska Hospital, Gothenburg, Gothenburg, Sweden
- Manchester University, Manchester, United Kingdom

REFERENCES:
- [Background] Barba E, Livovsky DM, Accarino A, Azpiroz F. Thoracoabdominal Wall Motion-Guided Biofeedback Treatment of Abdominal Distention: A Randomized Placebo-Controlled Trial. Gastroenterology. 2024 Aug;167(3):538-546.e1. doi: 10.1053/j.gastro.2024.03.005. Epub 2024 Mar 11. PMID 38467383
- [Result] Barba E, Accarino A, Azpiroz F. Correction of Abdominal Distention by Biofeedback-Guided Control of Abdominothoracic Muscular Activity in a Randomized, Placebo-Controlled Trial. Clin Gastroenterol Hepatol. 2017 Dec;15(12):1922-1929. doi: 10.1016/j.cgh.2017.06.052. Epub 2017 Jul 11. PMID 28705783